CLINICAL TRIAL: NCT06743802
Title: The Effect of Coenzyme Q10 in Preventing Pain After Thoracoscopic Surgery: a Randomized Controlled Trial
Brief Title: The Effect of Coenzyme Q10 in Preventing Pain After Thoracoscopic Surgery
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Coenzyme Q10 and pain
Record Dates: First submitted 2024-12-07; First posted 2024-12-20 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-11

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — coenzyme Q10

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Coenzyme Q10 (Experimental)
  Interventions: Drug: Coenzyme Q10
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Coenzyme Q10 — Coenzyme Q10 was administered from admission to one month after discharge at a dose of 200 mg per day (200 mg/qd).
  Arms: Coenzyme Q10
Other: Placebo — The placebo was administered from hospital admission until one month after discharge.
  Arms: Placebo

SUMMARY:
This study aimed to assess the effectiveness of Coenzyme Q10 in preventing both acute and chronic pain following thoracoscopic surgery, with a focus on its potential benefits in reducing the incidence and severity of pain.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75 years;
* American Society of Anesthesiology (ASA) physical status classification I-III;
* Scheduled for elective lung resection surgery under thoracoscopy;
* Voluntarily opting for patient-controlled intravenous analgesia;
* Willing to participate in this trial after consultation with the patient or their family and signing the informed consent form.

Exclusion Criteria:

* History of previous thoracotomy or thoracoscopic surgery;
* Patients converted to open thoracotomy intraoperatively;
* Severe hepatic or renal dysfunction;
* History of substance abuse;
* Pregnancy or breastfeeding;
* History of chronic pain;
* Use of coenzyme Q10 for more than one month;
* Allergy to coenzyme Q10;
* Patients unable to communicate or cooperate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
The incidence of chronic postsurgical pain | from the end of surgery to 3 months after surgery

SECONDARY OUTCOMES:
The incidence of acute postoperative pain with a score ≥4 | from the end of surgery to 6 hours,12 hours, 24 hours , 48 hours and 72 hours after surgery.
  Use pain Numeric Rating Scale(NRS) to evaluate the movement-evoked pain score and rest pain score. (NRS scale 0-10, where 0 was no pain, and 10 was the worst possible pain)
The severity of acute postoperative pain | from the end of surgery to 6 hours,12 hours, 24 hours , 48 hours and 72 hours after surgery.
  Use pain Numeric Rating Scale(NRS) to evaluate the movement-evoked pain score and rest pain score.(NRS scale 0-10, where 0 was no pain, and 10 was the worst possible pain)
The severity of chronic postsurgical pain | from the end of surgery to 3 months after surgery
  Use pain Numeric Rating Scale(NRS) to evaluate the movement-evoked pain score and rest pain score.(NRS scale 0-10, where 0 was no pain, and 10 was the worst possible pain)
The incidence of neuropathic pain | from the end of surgery to 3 months after surgery
  The DN4 questionnaire (Douleur Neuropathique 4) was used to evaluate neuropathic pain. The DN4 is a validated diagnostic tool consisting of 10 items, with scores ranging from 0 to 10. A score of 4 or higher indicates the presence of neuropathic pain.
The frequency of postoperative rescue analgesic use | from the end of surgery to 6 hours,12 hours, 24 hours , 48 hours and 72 hours after surgery.
The dose of analgesic use | from the end of surgery to 6 hours,12 hours, 24 hours and 48 hours after surgery.
The quality of recovery score at 3 days Postoperatively | from the end of surgery to 3 days.
  The QoR-15 scale, ranging from 0 to 150 with higher scores indicating better recovery, was used to assess the quality of recovery on postoperative day 3.
Health related quality of life score at 3 months Postoperatively | from the end of surgery to 3 months after surgery.
  The SF-8 scale, with a scoring range of 0 to 100 where higher scores indicate better physical and mental health, was used to evaluate health-related quality of life at 3 months postoperatively.
Postoperative length of hospital stay | from end of surgery to about 3 to 7 days after surgery.
The incidence of adverse reactions | From admission to 3 month post-discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Guangyou Duan, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Liu J, Li L, Luo L, Wu N, Xu F, Tao C, Chen J, Huang H, Duan G. Effect of coenzyme Q10 on pain prevention after thoracoscopic surgery: study protocol. Pain Manag. 2025 Dec;15(12):889-896. doi: 10.1080/17581869.2025.2567832. Epub 2025 Sep 30. PMID 41025845